CLINICAL TRIAL: NCT03312335
Title: Open-label, Monocentric, Phase II, Investigator-initiated Clinical Trial on Unbiased Characterization of Immunological Parameters in Interleukin-2-treated Systemic Lupus Erythematosus
Brief Title: Low-dose Interleukin-2 for Treatment of Systemic Lupus Erythematosus
Acronym: Charact-IL-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Onur Boyman, MD (Other)
Responsible Party: Sponsor-Investigator, Onur Boyman, MD, Professor and Chair, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: USZ-IM-001
Record Dates: First submitted 2017-09-29; First posted 2017-10-17 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Lupus Erythematosus, Systemic; SLE; Interleukin-2; IL-2; T-Lymphocytes, Regulatory; Treg
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low-dose Aldesleukin (Proleukin®) (Experimental)
  Interventions: Drug: Low-dose Aldesleukin (Proleukin®)

INTERVENTIONS:
Drug: Low-dose Aldesleukin (Proleukin®) — Subcutaneous injection of 1.5 million international units (MIU) of Aldesleukin (Proleukin®, Interleukin-2) once daily in 5-day courses every three weeks for a total of 4 cycles.

SUMMARY:
Systemic lupus erythematosus (SLE) is an autoimmune disease with multifactorial genesis. Recent research suggests a numerical and functional deficit of regulatory T (Treg) cells as an important contributing factor to the pathology seen in SLE. Treg cells play important roles in dampening overt stimulation of effector cells, as seen in many autoimmune diseases. As Treg cells are highly dependent on interleukin-2 (IL-2), application of low doses of IL-2 leads to markedly increased numbers and improved functionality of Treg cells in mice and humans. Several clinical trials investigated the safety of low-dose IL-2 treatment in different autoimmune diseases, including SLE. The trials conducted so far mainly focused on an increase in Treg cells after IL-2 treatment, not evaluating in detail the effects on other immune cells, presumably also playing important roles in the pathogenesis of SLE. For this reason, the investigators of this trial aim to conduct a complete phenotyping of cellular and soluble components in the blood of SLE patients treated with low-dose IL-2. Furthermore, the investigators want to offer this promising treatment to SLE patients in a controlled framework of an investigator initiated clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent forms as documented by signature.
* Diagnosis of SLE according to the criteria issued by the American College of Rheumatology.
* Female and male patients older than 18 years.
* Corticosteroids given at a stable dose for at least 4 weeks prior to enrollment.
* Immunosuppressive medication must be unchanged for at least 4 weeks prior to enrollment (e.g. mycophenolate-mofetil and/or methotrexate, see exclusion criteria).
* Participants must present with the following organ functions as defined below:
* Cardiac: No myocardial infarction prior to enrollment. No symptoms of heart failure New York Heart Association (NYHA) Class II or higher. No severe uncontrolled ventricular arrhythmias. No clinical signs of angina pectoris. No acute ischemia or active conduction system abnormalities additionally documented by an electrocardiogram prior to study enrollment.
* Pulmonary: forced expiratory volume 1 (FEV1) ≥50% (CTCAE grade 3 or lower) or diffusing capacity of the lungs for carbon monoxide (DLCO) ≥40% of predicted values.
* Renal: Glomerular filtration rate (GFR) ≥30 ml/min/1.73m2.
* Hepatic: Adequate hepatic function (aspartate aminotransferase [AST, also termed GOT] and alanine aminotransferase [ALT, also termed GPT] ≤2-fold upper limit of normal; total bilirubin <2.0 mg/dl, except for Gilbert-Meulengracht syndrome.
* The life expectancy of the patients should be greater than 12 months.

Exclusion Criteria:

* Contraindication to IL-2, e.g. known hypersensitivity or allergy.
* Solid organ transplant (allograft) recipient.
* Exposure to any new additional immunosuppressive medication within 4 weeks prior to enrollment.
* Exposure to rituximab 3 months prior to enrollment.
* Exposure to cyclophosphamide 3 months prior to enrollment.
* Following concomitant medications above the indicated maximal dose (given orally unless otherwise stated):

  g) Hydroxychloroquine, >400 mg/day h) Prednisone, >20 mg/day (or equivalent) i) Azathioprine, >2.5 mg/kg/day j) Mycophenolate-mofetil, >3 g/day k) Methotrexate, injected subcutaneously, >20 mg applied once weekly l) Belimumab, given intravenously, after induction >10 mg/kg every 4 weeks (only 4 participants with Belimumab treatment will be recruited, after this recruitment goal is achieved, Belimumab at any dose becomes an exclusion criteria)
* Simultaneous use of Sirolimus and Tacrolimus at the same time. Either agent alone is allowed. (Risk of thrombotic microangiopathy in chronic graft-versus-host disease patients)
* Participation in another study with investigational drug within 100 days preceding and during the present study.
* History of thrombotic thrombocytopenic purpura, hemolytic-uremic syndrome or thrombotic microangiopathy.
* Any active uncontrolled infection.
* Women who are pregnant or breast feeding.
* Intention to become pregnant during the course of the study.
* Lack of safe contraception, defined as:

Female participants of childbearing potential, not using, not willing to use, and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices in addition to the use of condoms. Note that female participants who are surgically sterilized / hysterectomized or post-menopausal for longer than 2 years are not considered as being of childbearing potential.

Male participants are obliged to use condoms as well to inform their partner about the participation in this trial. In addition, the partner must use a save method of contraception as described above.

* Other clinically significant concomitant disease states (e.g. renal failure, hepatic dysfunction, cardiovascular disease, etc.).
* Known or suspected non-compliance, drug or alcohol abuse.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders or dementia of the participant.
* Previous enrolment in the current study.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.
* Chronic infections:

  * HIV-positive individuals (increased risk of severe infections).
  * Patients suffering from active hepatitis B or C are ineligible.
  * Patients suffering from active tuberculosis are ineligible. Patients with latent tuberculosis may be eligible if patient received adequate tuberculostatic treatment.
* Any reason at the discretion of the treating physician where treatment with the investigational drug could indicate a risk for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Assessment of increase in percentage of Treg cells | Comparison between baseline (visit 2, day 0) and week 9 (visit 9, day 68).
  The primary outcome of this study is an increase in percentage of Treg cells of total CD4+ T cells between visit 2 (baseline) and week 9 (visit 9) measured in the blood of SLE patients not receiving Belimumab treatment. Treg cells are defined as CD3+CD4+CD127loCD25hiFoxp3+ and total CD4+ T cells are defined as CD3+CD4+.

SECONDARY OUTCOMES:
Exploratory assessment of cellular immune cell subsets in the blood of SLE patients. | Comparison between baseline (visit 2, day 0), visit 3 (day 5), visit 4 (day 21), visit 5 (day 26), visit 6 (day 42), visit 7 (day 47), visit 8 (day 63), visit 9 (day 68), visit 10 (day 96) and visit 11 (day 124).
  Different immune cell subsets isolated from whole blood will be quantified. Immune cells of interest will include: T cell subsets, including effector and regulatory CD4 and CD8 T cells, B cells, natural killer cells, innate lymphoid cells, dendritic cells, monocytes/macrophages, as well as eosinophil, basophil and neutrophil granulocytes and their respective subtypes including premature stages.
Exploratory assessment of soluble cytokines in the blood of SLE patients. | Comparison between baseline (visit 2, day 0), visit 3 (day 5), visit 4 (day 21), visit 5 (day 26), visit 6 (day 42), visit 7 (day 47), visit 8 (day 63), visit 9 (day 68), visit 10 (day 96) and visit 11 (day 124).
  Quantification of cytokines in the blood will include: common gamma chain cytokines, pro-inflammatory cytokines and anti-inflammatory cytokines.
Exploratory assessment of soluble CD25 in the blood of SLE patients. | Comparison between baseline (visit 2, day 0), visit 3 (day 5), visit 4 (day 21), visit 5 (day 26), visit 6 (day 42), visit 7 (day 47), visit 8 (day 63), visit 9 (day 68), visit 10 (day 96) and visit 11 (day 124).
  Soluble CD25 will be quantified in the serum of SLE patients.
Exploratory assessment of antibodies in the blood of SLE patients. | Comparison between baseline (visit 2, day 0), visit 3 (day 5), visit 4 (day 21), visit 5 (day 26), visit 6 (day 42), visit 7 (day 47), visit 8 (day 63), visit 9 (day 68), visit 10 (day 96) and visit 11 (day 124).
  Specific and unspecific antibodies will be quantified. This measurement will include Immunglobulin subclasses (IgA, IgG, IgD, IgM and IgE), anti-dsDNA, antinuclear, anti-Sm and anti-C1q antibodies.
Exploratory assessment of complement activity in SLE patients. | Comparison between baseline (visit 2, day 0), visit 3 (day 5), visit 4 (day 21), visit 5 (day 26), visit 6 (day 42), visit 7 (day 47), visit 8 (day 63), visit 9 (day 68), visit 10 (day 96) and visit 11 (day 124).
  Activity of complete and classical complement pathways will be determined.
Assessment of immune cells with immunohistochemistry and immunofluorescence in skin biopsies (optional outcome) | Comparison between baseline (visit 2, day 0) and week 9 (visit 9, day 68).
  Skin biopsies will be optional and only taken from patients signing a separate consent form.
Clinical response measured by the SELENA-SLEDAI score. | Comparison between baseline (visit 2, day 0), visit 5 (day 26), visit 9 (day 68) and visit 11 (day 124).
Clinical response measured by the BILAG-2004 score. | Comparison between baseline (visit 2, day 0), visit 5 (day 26), visit 9 (day 68) and visit 11 (day 124).
Clinical response measured by the Physician's Global Assessment (PGA) score. | Comparison between baseline (visit 2, day 0), visit 5 (day 26), visit 9 (day 68) and visit 11 (day 124).
Clinical response measured by the SLE Responder Index (SRI). | Comparison between baseline (visit 2, day 0), visit 5 (day 26), visit 9 (day 68) and visit 11 (day 124).
Reduction in dosing of concomitant medication. | Comparison between baseline (visit 2, day 0), visit 3 (day 5), visit 4 (day 21), visit 5 (day 26), visit 6 (day 42), visit 7 (day 47), visit 8 (day 63), visit 9 (day 68), visit 10 (day 96) and visit 11 (day 124).

OTHER OUTCOMES:
Incidence of adverse events (safety and tolerability) | Visit 2 (day 0), visit 3 (day 5), visit 4 (day 21), visit 5 (day 26), visit 6 (day 42), visit 7 (day 47), visit 8 (day 63), visit 9 (day 68), visit 10 (day 96) and visit 11 (day 124).
  Assessment of safety will be conducted by reporting adverse events. Frequency, severity and relation to IL-2 treatment will be evaluated and thoroughly described in the final report. Reporting will follow the Common Terminology Criteria for Adverse Events (CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: Onur Boyman, MD, Principal Investigator — Department of Immunology, University Hospital Zurich, University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided